CLINICAL TRIAL: NCT01145690
Title: Five Year Follow-up of Internet-based Cognitive Behaviour Therapy for Social Anxiety Disorder
Brief Title: Five Year Follow-up of Internet-based Cognitive Behaviour Therapy (CBT) for Social Anxiety Disorder (SAD)
Acronym: SOFIE-5YFU
Status: Completed | Type: Observational
Sponsor: Karolinska Institutet (Other)
Responsible Party: Nils Lindefors, MD, PHD, professor, Stockholm County Council and Karolinska Institute
Other Study IDs: SOFIE-5YFU
Record Dates: First submitted 2010-06-15; First posted 2010-06-17 (Estimated); Last update posted 2010-10-26 (Estimated); Status verified 2010-06

CONDITIONS: Social Anxiety Disorder
Keywords: cognitive behaviour therapy
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Internet-based CBT: All participants in this cohort received Internet-based CBT for social anxiety disorder in 2005. All participants were Swedish adults with a DSM-IV diagnosis of social anxiety disorder.

SUMMARY:
Social anxiety disorder (SAD) is one of the most prevalent anxiety disorders in the western world. Cognitive behavioural therapy (CBT) is the psychological treatment that has the largest empirical support. However, the availability to CBT is very limited in Sweden due to lack of therapists with proper training. Therefore it is important to evaluate alternative forms of treatment that are more time efficient. One of these methods is Internet based self-help therapy, which has proven to be an effective treatment for social anxiety disorder.

In this study, the investigators aim to conduct a follow-up assessment five years after completed Internet-based CBT. Participants received treatment within the context of a randomised controlled trial conducted in 2005. Thus, in the present study there will be no treatment interventions, only assessment.

ELIGIBILITY:
Inclusion Criteria:

* Must have a primary diagnosis of social phobia

Exclusion Criteria:

* Substance abuse during the last 6 months
* Other dominating diagnosis (not phobic personality disorder)
* A history of bipolar disorder or psychosis
* Major depression according to DSM-IV and >20 on madrs-s
* Risk of suicide
* Start of medication or change of dosis during the last 2 months
* Other parallel psychological treatment
* Previous CBT (last 3 years) for social phobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample is constituted by all 80 participants who received Internet-based CBT in 2005 within the context of a RCT in Sweden.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Measure of social anxiety and avoidance - Liebowitz Social Anxiety Scale (LSAS) | 5-year follow-up

SECONDARY OUTCOMES:
Measures of social anxiety in interaction and performance situations - SIAS & SPS | 5-year follow-up
Measure of depressive symptoms - MADRS-S | 5-year follow-up
Measure of general anxiety - BAI | 5-year follow-up
Measure of quality of life - QOLI | 5-year follow-up
Measure of social anxiety disorder diagnosis - SPSQ | 5-year follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Psykiatri Sydväst, Stockholm County Council, Stockholm, Stockholm County, Sweden

REFERENCES:
- [Derived] Hedman E, Furmark T, Carlbring P, Ljotsson B, Ruck C, Lindefors N, Andersson G. A 5-Year follow-up of internet-based cognitive behavior therapy for social anxiety disorder. J Med Internet Res. 2011 Jun 15;13(2):e39. doi: 10.2196/jmir.1776. PMID 21676694